CLINICAL TRIAL: NCT01099124
Title: Single-center, Open Trail of Phase 1 of M2ES With TC Regimen in Advanced NSCLC
Brief Title: Study of M2ES With Paclitaxel/Carboplatin (TC Regimen) in Advanced Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-CIH-CTI-001
Record Dates: First submitted 2010-02-24; First posted 2010-04-06 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2010-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: M2ES; NSCLC; Phase I Trial; Advanced NSCLC; Recurrent NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- M2ES combined with chemotherapy (Experimental)
  Interventions: Drug: M2ES

INTERVENTIONS:
Drug: M2ES — polyethylene glycol rh recombinant endostatin

SUMMARY:
The purpose of this study is to evaluate safety and tolerance of M2ES with TC regimen in advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years old;
2. Patients with Ⅲ/Ⅳ NSCLC confirmed by histopathology or cytology who ware naive or previous chemotherapy without TC regimen;
3. No contraindication for chemotherapy;
4. ECOG performance scale 0-2;
5. No history of anti-angiogenesis therapy;
6. Patients are voluntary to participate and sigh the informed contents.

Exclusion Criteria:

1. Concurrent use of other anti-cancer agents;
2. Allergic history to M2ES and biological agents;
3. Pregnant or breast-feeding women;
4. With other malignancy;
5. With severe cardiopulmonary disease;
6. Uncontrolled brain metastasis patients;
7. Other conditions that are regarded for exclusion by the trialists.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Adverse events incidence,including severe adverse events incidence | one year

SECONDARY OUTCOMES:
Tumor response rate and disease controlled rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kai LI, Principal Investigator — Tianjin Medical University Cancer Institude and Hospital
Locations (1):
- Tianjin Medical University Cancer Institude and Hospital, Tianjin, China